CLINICAL TRIAL: NCT05143398
Title: Effectiveness of a Rehabilitation Program (Nutritional + Physical Activity) in Sarcopenic Obesity
Brief Title: Nutritional Supplementation in Sarcopenic Obesity
Acronym: SARCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Amelia Brunani, Director of Clinical Unit, Istituto Auxologico Italiano
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018_06_28_05
Record Dates: First submitted 2021-11-10; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Sarcopenic Obesity
MeSH Terms: interventions — Diet; Proteins; Excitatory Amino Acids

STUDY DESIGN:
Intervention Model Description: After 1 week of standard diet (1650kcal/day with 18% protein) without physical activity, patients will be randomized into one of the 4 arms described below (20 subjects per study arm): 1st arm: low-calorie diet normoproteic with an energy deficit of 15% compared to what emerged from the calorimetric value (basal REE); 2nd arm: low-calorie diet normoproteic + an integration of 8.72 g of protein in the form of a nutritional supplement (18-20% protein; 3rd diet: low-calorie diet normoproteic + amino acid supplement (2 sachet/daily; 1 sachet contains protein 0 gr, carbohydrates 6.69 gr , lipids 0 gr, i-leucine 1,2 gr, i-isoleucine 0,6 gr, i-valine 0,6 gr). 4th diet: low-calorie diet normoproteic + an amino acid supplement (2 stick/daily; 1 stick pack contains protein 0 gr, carbohydrates 1,046 gr, lipids 0.074 gr, i-leucine 1.2 gr, i-isoleucine 0.6 gr, i-valine 0.6 gr, citric acid, succinic acid and malic acid). All patients perform daily aerobic physical activity/5 days/week for 4 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Diet Arm (Active Comparator): low-calorie diet normoproteic with an energy deficit of 15% compared to what emerged from the calorimetric value (basal REE)
  Interventions: Other: Diet
- Protein Arm (Active Comparator): low-calorie diet normoproteic + an integration of 8.72 g of protein in the form of a nutritional supplement (18-20% protein)
  Interventions: Dietary Supplement: Diet + protein
- EAA Arm (Active Comparator): low-calorie diet normoproteic + amino acid supplement (2 sachet/daily; 1 sachet contains protein 0 gr, carbohydrates 6.69 gr , lipids 0 gr, i-leucine 1,2 gr, i-isoleucine 0,6 gr, i-valine 0,6 gr).
  Interventions: Dietary Supplement: Diet + EAA
- EAA + TCA (Active Comparator): low-calorie diet normoproteic + an amino acid supplement (2 stick/daily; 1 stick pack contains protein 0 gr, carbohydrates 1,046 gr, lipids 0.074 gr, i-leucine 1.2 gr, i-isoleucine 0.6 gr, i-valine 0.6 gr, citric acid, succinic acid and malic acid)
  Interventions: Dietary Supplement: Diet + EAA and TCA

INTERVENTIONS:
Dietary Supplement: Diet + protein — Comparison of the efficacy
  Arms: Protein Arm
Dietary Supplement: Diet + EAA — Comparison of the efficacy
  Arms: EAA Arm
Dietary Supplement: Diet + EAA and TCA — Comparison of the efficacy
  Arms: EAA + TCA
Other: Diet — Comparison of the efficacy
  Arms: Diet Arm

SUMMARY:
The obese patient presents a quantitative and qualitative deficit of muscle mass as occurs in the elderly subject that was named Sarcopenic Obesity (SO). The use of a diet that includes protein supplements and / or essential amino acids seems to improve this condition in the elderly; there are no similar studies in obese subjects, in particular during a low-calorie diet and physical activity program that can produce further loss of muscle mass. This study aims to verify whether the administration of these supplements (protein or amino acid) in the obese patient are effective in improving anthropometric and functional parameters and some serum markers of muscle metabolism. The results obtained could represent new therapeutic protocols in the treatment of obesity.

DETAILED DESCRIPTION:
Several studies have confirmed that adequate nutrition, especially protein intake, including at breakfast, or supplementation with amino acids, in association with adequate physical activity plays an important role in the treatment of SO.

The supplementation of protein or amino acid preparations (in particular with the 9 essential amino acids including, the branched - leucine, isoleucine, valine), marketed in different formulations, has already allowed to document a significant therapeutic efficacy in the treatment of elderly sarcopenic subjects. In fact, the use of these preparations improves physical performance and muscle strength by inducing the synthesis of proteins involved in the biogenesis and functionality of mitochondria - that is, the cellular organelles responsible for the production of energy in the form of ATP - and of myofibrillar proteins (which constitute the large percentage of muscle mass), both in laboratory animals and in humans.

ELIGIBILITY:
Inclusion Criteria:

* patients with obesity (BMI> 35kg / m2)
* sarcopenia (criteria described in Coltorti A et al).

Exclusion Criteria:

* renal insufficiency
* diabetes
* muscular pathologies
* neurological-neurodegenerative pathologies
* cognitive decline

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Change of Body weight | basal and at 4 weeks
  weight in kilograms
Change of Height | basal and at 4 weeks
  height in meters
Change of BMI | basal and at 4 weeks
  weight and height will be combined to report BMI in kg/m^2
Change of Waist | basal and at 4 weeks
  waist circumference in centimeters
Change of FM | basal and at 4 weeks
  Fat Mass (FM) in % of body weight in kilograms
Change of FFM | basal and at 4 weeks
  Free Fat Mass (FFM) in % of body weight in kilograms
Change of MM | basal and at 4 weeks
  Muscle Mass (MM) in % of body weight in kilograms
Change of Muscle strenght | basal and at 4 weeks
  muscle streght at the hand (right and left) in kg
Change of Walking | basal and at 4 weeks
  6 minute walk test (6MWT), meters walking in 6 minutes
Change of TUG | basal and at 4 weeks
  time, in second, to up from the chair, walks 3 meters, turns around, walks back to the chair and sits down
Change of Metabolic profile | basal and at 4 weeks
  glycaemia, total cholesterol, LDL cholesterol, triglycerides all in mg/dl
Change of Insulin secretion | basal and at 4 weeks
  insulin pasma levels in mU/l
Change of Homa index | basal and at 4 weeks
  glycaemia and insulin will be combined to report Homa index in mmol/l/mU/l
Change of Muscle function | basal and at 4 weeks
  irisin and procollagen type III N-terminal peptide (P3NP) in ng/ml
Change of Muscle wasting | basal and at 4 weeks
  C-terminal agrin fragment (CAF) in pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Brunani, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- Amelia Brunani, Verbania, VB, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsu KJ, Liao CD, Tsai MW, Chen CN. Effects of Exercise and Nutritional Intervention on Body Composition, Metabolic Health, and Physical Performance in Adults with Sarcopenic Obesity: A Meta-Analysis. Nutrients. 2019 Sep 9;11(9):2163. doi: 10.3390/nu11092163. PMID 31505890
- [Background] Wang X, Miller GD, Messier SP, Nicklas BJ. Knee strength maintained despite loss of lean body mass during weight loss in older obese adults with knee osteoarthritis. J Gerontol A Biol Sci Med Sci. 2007 Aug;62(8):866-71. doi: 10.1093/gerona/62.8.866. PMID 17702878
- [Background] Frimel TN, Sinacore DR, Villareal DT. Exercise attenuates the weight-loss-induced reduction in muscle mass in frail obese older adults. Med Sci Sports Exerc. 2008 Jul;40(7):1213-9. doi: 10.1249/MSS.0b013e31816a85ce. PMID 18580399
- [Background] Malafarina V, Uriz-Otano F, Malafarina C, Martinez JA, Zulet MA. Effectiveness of nutritional supplementation on sarcopenia and recovery in hip fracture patients. A multi-centre randomized trial. Maturitas. 2017 Jul;101:42-50. doi: 10.1016/j.maturitas.2017.04.010. Epub 2017 Apr 22. PMID 28539168
- [Background] Rondanelli M, Opizzi A, Antoniello N, Boschi F, Iadarola P, Pasini E, Aquilani R, Dioguardi FS. Effect of essential amino acid supplementation on quality of life, amino acid profile and strength in institutionalized elderly patients. Clin Nutr. 2011 Oct;30(5):571-7. doi: 10.1016/j.clnu.2011.04.005. Epub 2011 Jun 1. PMID 21636183
- [Background] D'Antona G, Ragni M, Cardile A, Tedesco L, Dossena M, Bruttini F, Caliaro F, Corsetti G, Bottinelli R, Carruba MO, Valerio A, Nisoli E. Branched-chain amino acid supplementation promotes survival and supports cardiac and skeletal muscle mitochondrial biogenesis in middle-aged mice. Cell Metab. 2010 Oct 6;12(4):362-372. doi: 10.1016/j.cmet.2010.08.016. PMID 20889128
- [Background] Solerte SB, Gazzaruso C, Bonacasa R, Rondanelli M, Zamboni M, Basso C, Locatelli E, Schifino N, Giustina A, Fioravanti M. Nutritional supplements with oral amino acid mixtures increases whole-body lean mass and insulin sensitivity in elderly subjects with sarcopenia. Am J Cardiol. 2008 Jun 2;101(11A):69E-77E. doi: 10.1016/j.amjcard.2008.03.004. PMID 18514630
- [Background] Valerio A, D'Antona G, Nisoli E. Branched-chain amino acids, mitochondrial biogenesis, and healthspan: an evolutionary perspective. Aging (Albany NY). 2011 May;3(5):464-78. doi: 10.18632/aging.100322. PMID 21566257
- [Background] Coltorti A, Scalfi L, Borrelli R, Contaldo F, Diaz E. [Validity of 5 bioelectric impedance equations for the estimation of lean body mass in women]. Minerva Endocrinol. 1991 Jan-Mar;16(1):37-41. Italian. PMID 1944015
- [Derived] Brunani A, Cancello R, Gobbi M, Lucchetti E, Di Guglielmo G, Maestrini S, Cattaldo S, Pitera P, Ruocco C, Milesi A, Valerio A, Capodaglio P, Nisoli E. Comparison of Protein- or Amino Acid-Based Supplements in the Rehabilitation of Men with Severe Obesity: A Randomized Controlled Pilot Study. J Clin Med. 2023 Jun 25;12(13):4257. doi: 10.3390/jcm12134257. PMID 37445292